CLINICAL TRIAL: NCT03959098
Title: Observational Study on Effectiveness and Safety of Integrative Korean Medicine Treatment for Cervical Disc Herniation With Radiculopathy
Brief Title: Effectiveness and Safety of Korean Medicine Treatment for Cervical Disc Herniation
Status: Active, not recruiting | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, K.M.D, Rehabilitation Medicine Specialist, Jaseng Medical Foundation
Other Study IDs: JS-CT-2019-02
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain; Cervical Radiculopathy; Intervertebral Disc Displacement
Keywords: Korean Medicine; Effectiveness; Neck Pain
MeSH Terms: conditions — Neck Pain; Radiculopathy; Intervertebral Disc Displacement | interventions — Phytotherapy; Acupuncture Therapy; Electroacupuncture; Cupping Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine will be administered in water-based decoction (120ml) and dried powder (2g) form (Ostericum koreanum,Eucommia ulmoides, canthopanax sessiliflorus, Achyranthes japonica, Psoralea corylifolia, aposhnikovia divaricata, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, Glycinemax, Atractylodes japonica) at the physician's discretion.
  Other Names: Traditional herbal medicine
Procedure: Chuna manual medicine — Chuna is a Korean manual therapy directed at the spine and joints that incorporates various spinal manual medicine techniques for joint mobilization involving highvelocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement. Chuna manual medicine will be administered to the pelvic, lumbar, thoracic, and cervical vertebrae at the physician's discretion.
  Other Names: Chuna manipulation
Procedure: Bee venom pharmacopuncture — Bee venom pharmacopuncture will be administered only after confirming a negative response to hypersensitivity skin test. Diluted bee venom saline:bee venom ratio, 10,000:1) filtered for allergens will usually be injected at 4-5 acupoints proximal to the dysfunctional site at the physician's discretion. Each acupuncture point will be injected to a total of 0.5-1 cc using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, hinchang medical co., Korea).
  Other Names: Bee venom acupuncture
Procedure: Pharmacopuncture — Pharmacopuncture consisting of select herbal ingredients will be dministered at Hyeopcheok (Huatuo Jiaji, EX B2), Ah-shi points and local acupuncture points using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea) at the physician's discretion.
Procedure: Acupuncture — Acupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Electroacupuncture — Electroacupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Cupping — Cupping treatment will be administered at 1-2 points using mainly proximal acupuncture points and Ah-shi points.
Procedure: Other intervention(s) — Patients will be allowed any other additional intervention(s) as deemed necessary regardless of type or dose, and patterns of use will be investigated and recorded as a pragmatic clinical study.

SUMMARY:
A prospective observational study investigating the effectiveness and safety of integrative Korean medicine treatment in cervical disc herniation patients with neck pain or cervical radiculopathy at 4 locations of Jaseng Hospital of Korean Medicine as assessed through of pain, functional disability, work loss and quality of life patient-reported outcomes

DETAILED DESCRIPTION:
This is a prospective observational study to the aim of investigating the effectiveness and safety of integrative Korean medicine treatment (generally consisting of herbal medicine, Chuna manual medicine, bee venom pharmacopuncture and pharmacopuncture, acupuncture, electroacupuncture, and cupping) in cervical disc herniation patients with neck pain or cervical radiculitis diagnosed by cervical MRI and clinical symptoms including cervical radiculopathy at 4 locations of Jaseng Hospital of Korean Medicine (Gangnam, Bucheon, Daejeon, Haeundae) as assessed through of pain, functional disability, work loss, and quality of life patient-reported outcomes with a 5-year follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 19 years ~ 65 years
* Patients with one arm pain or both side arm pain or neck pain with intensity of NRS ≥6 which occurred less then 12 month before
* Patients with cervical radiculopathy symptoms of one or both side of arms
* Patients diagnosed with cervical disc herniation with over protrusion degree of prolapsed inter-vertebral disc assessed on MRI
* Patients with plans of receiving Korean medicine treatment for cervical disc herniation for ≥2 months
* Patients who have agreed to study participation

Exclusion Criteria:

* Patients with other systemic diseases that may interfere with treatment effect or outcome interpretation
* Patients with soft tissue pathologies or pathologies of non-spinal origin that may cause neck pain or radiating arm pain (e.g. spinal tumor, rheumatoid arthritis)
* Patients with medical history of cervical myelopathy which can cause neck pain or radiating arm pain
* Patients with medical history of surgery in relation with cervical disc herniation
* Patients for whom acupuncture treatment may be inappropriate or unsafe (e.g. hemorrhagic diseases, blood clotting disorders, history of anticoagulation medicine intake, serious diabetes with risk of infection, severe cardiovascular diseases, or other conditions deemed unsuitable for acupuncture treatment)
* Pregnant patients or patients planning pregnancy
* Patients with serious psychological disorders
* Patients unable to fill out study participation consent form
* Patients deemed unsuitable for study participation as assessed by the researchers

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms of neck pain or radiating arm pain alongside cervical radiculopathy symptoms
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Numeric rating scale (NRS) out of neck pain and radiating arm pain | Time Frame: Change from baseline to 4 months
  Change from higher score at baseline out of neck pain or radiating arm pain intensity to same score at 4 months. Total score range: -10 (worse outcome) to 10 (better outcome) Total score range: -10 (worse outcome) to 10 (better outcome)

SECONDARY OUTCOMES:
Visual analogue scale (VAS) of neck pain | Time Frame: Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Neck pain intensity for the past 3 days. Total score range: 0 (better outcome) to 100 (worse outcome)
Visual analogue scale (VAS) of radiating arm pain | Time Frame: Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Radiating arm pain intensity for the past 3 days. Total score range: 0 (better outcome) to 100 (worse outcome)
Neck Disability Index (NDI) | Time Frame: Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range: 0 (better outcome) to 50 (worse outcome)
Patient Global Impression of Change (PGIC) | Time Frame: 8, 16, 20, 24 weeks, 1, 3, 5 years
  Global patient-reported outcome. Total score range: 1 (better outcome) to 7 (worse outcome)
EuroQol 5-dimensions 5-levels (EQ-5D-5L) | Time Frame: Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Health-related quality of life questionnaire. Total score range: 11111 (better outcome) to 55555 (worse outcome)
Type and frequency of other intervention(s) | Baseline, 4, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Use of any other additional intervention(s) other than the integrative Korean medicine treatment administered by the attending physician (start date of treatment, end date of treatment, name of treatment, number of treatment sessions received, and other comments)
Physical examination | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Cervical physical examination
Type and frequency of adverse reaction(s) | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Safety
Numeric rating scale (NRS) of Neck pain | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Neck pain intensity for the past 3 days. Total score range: 0 (better outcome) to 10 (worse outcome)
Numeric rating scale (NRS) of radiating arm pain | Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  Radiating arm pain intensity for the past 3 days. Total score range: 0 (better outcome) to 10 (worse outcome)
SF-36 | Baseline, 4, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
EQ-VAS | [Time Frame: Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks, 1, 3, 5 years]
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.

CONTACTS AND LOCATIONS:
Overall Officials: Won-Il Ko, KMD, Principal Investigator — Jaseng Hospital of Korean Medicine; Sun-A Kim, KMD, Principal Investigator — Daejeon Jaseng Hospital of Korean Medicine; Hyun-Woo Cho, KMD, Principal Investigator — Haeundae Jaseng Hospital of Korean Medicine; Ji-Yun Seo, KMD, Principal Investigator — Bucheon Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Medical Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No